CLINICAL TRIAL: NCT00185939
Title: The Use of Prophylactic Antibiotics In the Management of Dog Bites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: K23AR002137 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Bite; Wound; Infection
Keywords: dog bites; infection; prophylactic antibiotics; cost effectiveness
MeSH Terms: conditions — Bites and Stings; Wounds and Injuries; Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Augmentin

SUMMARY:
This double blinded RCT will help to ascertain the usefulness of prophylactic antibiotics in the management of uncomplicated dog bites, utilizing currently best available antibiotics (Augmentin) and an important clinical outcome of infection.

By enrolling 100-150 patients in this pilot trial as part of a k-award the investigators plan to utilize the point estimates of infection, side effects and other important outcomes and incorporate these into a cost most to determine the most cost effective management of these wounds and to determine if further study is warranted based on the findings.

DETAILED DESCRIPTION:
This double blinded RCT will help to ascertain the usefulness of prophylactic antibiotics in the management of uncomplicated dog bites, utilizing currently best available antibiotics (Augmentin) and an important clinical outcome of infection.

By enrolling 100-150 patients in this pilot trial as part of a k-award the investigators plan to utilize the point estimates of infection, side effects and other important outcomes and incorporate these into a cost most to determine the most cost effective management of these wounds and to determine if further study is warranted based on the findings.

ELIGIBILITY:
Inclusion Criteria:

All patients including all children and English speaking/reading persons who present with a full thickness dog bite to participating emergency departments will be considered. Non-English speaking/reading subjects for whom we can provide translation for will also be considered.

Exclusion Criteria:

Exclusion Criteria:

* allergy to penicillin or amoxicillin/clavulanic acid
* wounds presenting with an active infection (require antibiotics) or greater than 12 hours old.
* patients with underlying fracture, joint or neurovascular injury, or multiple trauma requiring specialty referral. Specifically any broken skin over a joint will need treatment and be excluded from the study and randomization.
* patients on immunosuppressive agents, prolonged chronic steroid use (defined as continuous use for > 14 days, 3 times a year) active HIV disease (determined by treating physician on history) or splenectomized. (could skew one group and at risk for overwhelming sepsis and death if infected)
* patients unwilling or unable to complete the required follow-up, and those unable to provide a contact phone number

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125
Dates: Start 2003-08; Study Completion 2005-11

PRIMARY OUTCOMES:
Wound infection

SECONDARY OUTCOMES:
side effects of medication

CONTACTS AND LOCATIONS:
Overall Officials: James V Quinn, MD MS, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Mills Peninsula Hospital, Burlingame, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California